CLINICAL TRIAL: NCT07030543
Title: Feasibility Of Individualized Dietary Plan (Idp) On Glycemic Control And Total Cholestrol In Diabetic Patients At Diabetes Hospital And Research Centre Peshawar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr Khalid Rahman, Director IPHSS, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/016
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Glycemic Control; Cardiovascular Risk Factors; Individualized Dietary Plan (IDP)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Inosine Diphosphate; Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized, open-label feasibility trial with two arms: an intervention group receiving individualized dietary plans (IDPs) and a control group receiving standard dietary advice. Participants (n=122) will be randomly assigned using simple random sampling, with no masking (open-label) due to the nature of dietary interventions. The study will assess feasibility through adherence (PDAQ scores) and acceptability (recruitment rates), while secondary outcomes include changes in HbA1c, cholesterol, and BMI over 3 months. The design ensures practical evaluation of IDPs in a real-world clinical setting at Diabetes Hospital Peshawar.
Masking Description: This is an open-label study with no masking (blinding) of participants, care providers, investigators, or outcomes assessors. The nature of the dietary intervention makes blinding impractical, as both the individualized meal plans and standard advice require active participation and awareness from patients and providers. However, objective laboratory measures (HbA1c, cholesterol) will be used to minimize bias in outcome assessment. The study acknowledges potential performance bias due to the lack of masking but prioritizes real-world applicability in evaluating the feasibility of personalized nutrition for diabetes management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Dietary Plan (IDP) Group (Experimental): Participants in this arm will receive a personalized dietary plan (IDP) tailored by a dietitian based on their BMI, glycemic levels, age, and lifestyle. The IDP includes Low-glycemic index foods (lentils, whole grains, barley), High-fiber foods (vegetables, cereals), Healthy fats (fish, walnuts, olive oil), Restricted high-sugar foods (rice, potatoes) and saturated fats (fried foods), Adherence will be monitored weekly using the Perceived Dietary Adherence Questionnaire (PDAQ) over 10 weeks.
  Interventions: Behavioral: Individualized Dietary Plan (IDP) for Type 2 Diabetes
- Standard Care Group (Active Comparator): Participants will receive conventional dietary advice for diabetes management (non-personalized), as routinely provided at the Diabetes Hospital and Research Centre Peshawar. This includes general guidelines on carbohydrate intake, portion control, and avoidance of sugary foods, without individualized adjustments.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Individualized Dietary Plan (IDP) for Type 2 Diabetes — This study evaluates the feasibility of an Individualized Dietary Plan (IDP), a structured, patient-tailored nutrition intervention designed to improve glycemic control and lipid profiles in adults with Type 2 Diabetes Mellitus (T2DM).
  Other Names: Personalized Nutrition Therapy, Medical Nutrition Therapy (MNT), Diabetes-Specific Meal Plan
  Arms: Individualized Dietary Plan (IDP) Group
Behavioral: Usual care — Standard dietary advice as per the current clinical practice.
  Arms: Standard Care Group

SUMMARY:
This study aims to test whether a personalized meal plan (Individualized Dietary Plan, IDP) is practical and helpful for adults with type 2 diabetes in Peshawar, Pakistan. We want to see if patients can follow the IDP for 10 weeks and if it improves their blood sugar control and cholesterol levels. About 122 participants will be randomly assigned to either the IDP group (receiving customized diet advice) or a standard care group. We will measure their weight, blood sugar (HbA1c), cholesterol, and other health markers at the start and after 3 months. Results will show if a larger study is feasible in our local community.

DETAILED DESCRIPTION:
Type 2 diabetes prevalence in Pakistan is high (16.98%), yet standardized dietary advice is often given without considering individual factors like age, weight, or lifestyle. Evidence shows nutrition therapy improves glycemic control, but no studies have tested personalized dietary plans in Pakistan's local population. This feasibility trial addresses this gap by evaluating the practicality of implementing IDPs at the Diabetes Hospital and Research Centre Peshawar.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with physician-diagnosed Type 2 Diabetes Mellitus.
* Receiving care at Diabetes Hospital and Research Centre Peshawar.
* Willing to comply with dietary interventions and follow-up.

Exclusion Criteria:

* Pregnant women (to exclude gestational diabetes).
* Patients with conditions preventing dietary adherence (severe comorbidities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Adherence | Baseline to 3 months.
  Measures participant adherence to the IDP using the Perceived Dietary Adherence Questionnaire (PDAQ).
  The scoring of the questionnaire are as follows:
  Good Adherence: Score ≥70 (consistent adherence over 10 weeks).
  Poor Adherence: Score 45-69 (inconsistent adherence over 7-9 weeks).
Acceptability - Recruitment Rate | Enrollment to study completion (6 months)
  Assesses acceptability via recruitment rate, calculated as:
  Formula: (Number of participants completing 3 month follow-up) ÷ (Number of randomized participants) × 100.
Change in Glycemic Control (HbA1c) | Baseline to 3 months
  Measures difference in HbA1c levels (reflecting 3-month average blood glucose) between IDP and control groups.
  The threshold of glycemic control are as follows:
  Normal: <7%. Abnormal: ≥7%.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Naz, MPH, Principal Investigator — Khyber Medical Univeristy Peshawar
Locations (1):
- Diabetes Hospital and Research Centre, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study will be shared with qualified researchers to support reproducibility and further scientific inquiry. This includes:
  Baseline characteristics (age, sex, BMI, HbA1c, cholesterol levels)
  Adherence scores (PDAQ questionnaire results)
  Outcome measures (HbA1c, total cholesterol, fasting blood sugar at 3-month follow-up)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available 6 months after study completion (final publication).
  Shared data will remain accessible for 5 years via the repository.
Access Criteria: Data will be available to qualified researchers with a methodologically sound proposal approved by an independent review committee. Requestors must sign a data use agreement outlining ethical restrictions.

REFERENCES:
- [Background] Mottalib A, Salsberg V, Mohd-Yusof BN, Mohamed W, Carolan P, Pober DM, Mitri J, Hamdy O. Effects of nutrition therapy on HbA1c and cardiovascular disease risk factors in overweight and obese patients with type 2 diabetes. Nutr J. 2018 Apr 7;17(1):42. doi: 10.1186/s12937-018-0351-0. PMID 29626933
- [Background] Aamir AH, Ul-Haq Z, Mahar SA, Qureshi FM, Ahmad I, Jawa A, Sheikh A, Raza A, Fazid S, Jadoon Z, Ishtiaq O, Safdar N, Afridi H, Heald AH. Diabetes Prevalence Survey of Pakistan (DPS-PAK): prevalence of type 2 diabetes mellitus and prediabetes using HbA1c: a population-based survey from Pakistan. BMJ Open. 2019 Feb 21;9(2):e025300. doi: 10.1136/bmjopen-2018-025300. PMID 30796126
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228